CLINICAL TRIAL: NCT06021353
Title: Contralateral Study of the WaveLight® Ultraviolet Femtosecond Laser, Model 1026 Versus the WaveLight® FS200 Infrared Femtosecond Laser, Model 1025 for Corneal Flap Creation
Brief Title: Contralateral Study of WaveLight® Femtosecond Laser Devices for Corneal Flap Creation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFO268-E005
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UV fs-Laser (Other): First surgical eye randomly assigned to the UV fs-Laser with the second surgical eye (fellow eye) assigned to the IR fs-Laser for the purpose of corneal flap creation during LASIK surgery
  Interventions: Device: UV fs-Laser; Procedure: LASIK
- IR fs-Laser (Other): First surgical eye randomly assigned to the IR fs-Laser with the second surgical eye (fellow eye) assigned to the UV fs-Laser for the purpose of corneal flap creation during LASIK surgery
  Interventions: Device: IR fs-Laser; Procedure: LASIK

INTERVENTIONS:
Device: UV fs-Laser — Stationary scanning spot femtosecond laser used for corneal flap creation during refractive surgery
  Other Names: WaveLight Ultraviolet Femtosecond Laser Model 1026 with Patient Interface Model 1507
  Arms: UV fs-Laser
Device: IR fs-Laser — Stationary scanning spot femtosecond laser used for corneal flap creation during refractive surgery
  Other Names: WaveLight FS200 Infrared Femtosecond Laser Model 1025 with Patient Interface Model 1515
  Arms: IR fs-Laser
Procedure: LASIK — Laser-assisted in situ keratomileusis (LASIK) surgery

SUMMARY:
The purpose of this study is to assess the WaveLight Ultraviolet Femtosecond Laser System, Model 1026 (UV fs-Laser) corneal flap creation accuracy as compared to the already marketed WaveLight FS200 Infrared Femtosecond Laser, Model 1025 (IR fs-Laser).

DETAILED DESCRIPTION:
Subjects who qualify to participate will have both eyes treated in the study (one eye with the UV fs-Laser and the other eye with the IR fs-Laser) and will attend a total of 5 study visits over a period of approximately 2 months. This study will be conducted outside the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Good ocular health;
* Natural lens with no evidence of cataract;
* Eligible for LASIK;
* Stable refraction;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Presence of dry eye;
* Contraindicated systemic disease or ocular conditions;
* Treatment with a contraindicated medication;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum deviation of corneal flap thickness at the margins from achieved central flap thickness at 1 month | Month 1
  Corneal flap thickness will be measured using optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Clinical Trial Lead, CRD Surgical, Study Director — Alcon Research, LLC
Locations (1):
- Personaleyes, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No